CLINICAL TRIAL: NCT04290988
Title: Circuitry Assessment and Reinforcement Training Effects on Recovery (CARTER)
Brief Title: Circuitry Assessment and Reinforcement Training Effects on Recovery
Acronym: CARTER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00242136
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Aphasia; Primary Progressive Aphasia; Stroke
Keywords: communication; language; speech; anxiety; sleep; neurofeedback
MeSH Terms: conditions — Aphasia; Aphasia, Primary Progressive; Stroke; Communication; Language; Speech; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: To evaluate the effects of EEG neurofeedback on communication skills in participants with post-stroke aphasia and primary progressive aphasia (PPA), this study will utilize a randomized double-blind, sham-controlled, within-subject crossover trial design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active EEG Neurofeedback (Experimental): 15 sessions of active EEG neurofeedback at a frequency of 3-5 sessions per week for a duration of 3-5 weeks.
  Interventions: Device: EEG Neurofeedback
- Sham Feedback (Sham Comparator): 15 sessions of sham neurofeedback at a frequency of 3-5 sessions per week for a duration of 3-5 weeks.
  Interventions: Device: Sham Feedback

INTERVENTIONS:
Device: EEG Neurofeedback — Active EEG neurofeedback
  Arms: Active EEG Neurofeedback
Device: Sham Feedback — Sham EEG feedback sessions identical to active sessions except that the feedback given to the participant will not be based on the individual's live EEG activity.
  Arms: Sham Feedback

SUMMARY:
This study investigates if electroencephalography (EEG) neurofeedback training is more beneficial than sham feedback training for the improvement of communication, anxiety, and sleep quality in individuals with aphasia. Half of the participants will receive active EEG neurofeedback sessions first, followed by sham feedback sessions in a crossover design. The other half of participants will undergo sham feedback sessions first, followed by active neurofeedback.

DETAILED DESCRIPTION:
Neurofeedback, a form of biofeedback, provides a visual and/or audio representation of an individual's neural electrical activity from live EEG recording. Using operant conditioning principles, individuals are trained to increase or reduce patterns of brainwave activity to modify behavior and performance. Although neurofeedback has not yet been investigated as a treatment for aphasia or other communication deficits due to stroke or neurodegenerative disease, it may be effective. Previous studies have observed improvement in cognitive and behavioral measures in those with conditions such as Attention Deficit Disorder and Attention Deficit Hyperactivity Disorder. Furthermore, it has been associated with reduced anxiety and sleep disruption, which both exacerbate language and communication impairments. Research is needed to determine if neurofeedback may be an effective treatment for language disorders such as PPA and post-stroke communication disorders.

It is possible that EEG neurofeedback, which focuses on improving abnormal brainwave patterns, could provide certain therapeutic benefits to individuals with PPA or post-stroke aphasia, either by directly affecting neural networks that underlie language, or more generally by reducing anxiety and inattention through behavioral conditioning. Reduction of anxiety in neurological diseases can be beneficial not only for functional performance but also sleep duration and quality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPA or aphasia secondary to stroke and presence of naming deficits with confirmation of diagnosis by neurologist
* Capable of giving informed consent or indicating another to provide informed consent
* Age 18 or older.
* If aphasia is secondary to stroke, the stroke must have occurred between 6 months and 5 years prior to enrollment in the study.

Exclusion Criteria:

* Lack of English proficiency
* Not medically stable
* Picture naming accuracy above 80% on the Philadelphia Naming Test (PNT)
* Prior history of neurologic disease affecting the brain (e.g., brain tumor, multiple sclerosis, traumatic brain injury) other than stroke or PPA and its underlying neurological pathologies: Alzheimer's Disease, Frontotemporal Lobar Degeneration or Dementia with Lewy bodies
* Prior history of severe psychiatric illness, developmental disorders or intellectual disability (e.g., PTSD, major depression, bipolar disorder, schizophrenia, obsessive compulsive disorder (OCD), autism spectrum disorders)
* Uncorrected severe visual loss or hearing loss by self-report and medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argye E Hillis, MD, MA, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banerjee S, Argaez C. Neurofeedback and Biofeedback for Mood and Anxiety Disorders: A Review of Clinical Effectiveness and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2017 Nov 13. Available from http://www.ncbi.nlm.nih.gov/books/NBK531603/ PMID 30299634
- [Background] Berube S, Nonnemacher J, Demsky C, Glenn S, Saxena S, Wright A, Tippett DC, Hillis AE. Stealing Cookies in the Twenty-First Century: Measures of Spoken Narrative in Healthy Versus Speakers With Aphasia. Am J Speech Lang Pathol. 2019 Mar 11;28(1S):321-329. doi: 10.1044/2018_AJSLP-17-0131. PMID 30242341
- [Background] Collura, T. (2014). Technical foundations of neurofeedback. New York: Taylor and Francis.
- [Background] Fuchs T, Birbaumer N, Lutzenberger W, Gruzelier JH, Kaiser J. Neurofeedback treatment for attention-deficit/hyperactivity disorder in children: a comparison with methylphenidate. Appl Psychophysiol Biofeedback. 2003 Mar;28(1):1-12. doi: 10.1023/a:1022353731579. PMID 12737092
- [Background] Hetkamp M, Bender J, Rheindorf N, Kowalski A, Lindner M, Knispel S, Beckmann M, Tagay S, Teufel M. A Systematic Review of the Effect of Neurofeedback in Cancer Patients. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419832361. doi: 10.1177/1534735419832361. PMID 30832518
- [Background] Nan W, Dias APB, Rosa AC. Neurofeedback Training for Cognitive and Motor Function Rehabilitation in Chronic Stroke: Two Case Reports. Front Neurol. 2019 Jul 24;10:800. doi: 10.3389/fneur.2019.00800. eCollection 2019. PMID 31396152
- [Background] Wang SY, Lin IM, Fan SY, Tsai YC, Yen CF, Yeh YC, Huang MF, Lee Y, Chiu NM, Hung CF, Wang PW, Liu TL, Lin HC. The effects of alpha asymmetry and high-beta down-training neurofeedback for patients with the major depressive disorder and anxiety symptoms. J Affect Disord. 2019 Oct 1;257:287-296. doi: 10.1016/j.jad.2019.07.026. Epub 2019 Jul 5. PMID 31302517

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants were enrolled. 1 participant withdrew before randomization.
Groups:
- Active EEG Neurofeedback, Then Sham Neurofeedback: 15 sessions of active neurofeedback at a frequency of 3-5 sessions per week for a duration of 3-5 weeks followed by 15 sessions of sham neurofeedback at a frequency of 3-5 sessions per week for a duration of 3-5 weeks.
- Sham Feedback, Then Active Neurofeedback: 15 sessions of sham neurofeedback at a frequency of 3-5 sessions per week for a duration of 3-5 weeks followed by 15 sessions of active neurofeedback at a frequency of 3-5 sessions per week for a duration of 3-5 weeks.
Period: Overall Study
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (27.3) | 80 (3.5) | 67.3 (22.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Philadelphia Naming Test [Mean (Standard Deviation); unit: score on a scale] — The score range is 0 - 175 (higher scores reflect more accurate naming/better naming ability
  score on a scale | 59 (49.4) | 85 (74.7) | 72 (58.4)
Controlled Oral Word Association (COWA) [Mean (Standard Deviation); unit: score on a scale] — Score ranges from 0 to the total number of correct words that begin with one of the letters in the set. There is no ceiling of a maximum score. Higher numbers reflect better verbal fluency.
  score on a scale | 4 (4.6) | 7.5 (10.6) | 5.4 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Items Correctly Named on the Philadelphia Naming Test
Description: Change in number of items correctly named on a behavioral picture naming assessment. The score range is 0 - 175 (higher scores reflect more accurate naming/better naming ability)
Time Frame: Baseline, 1 week following each intervention period
Measure: Mean (Standard Deviation); unit: Number of Items Correct on Naming Test
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
Number of Items Correct on Naming Test
  Difference Post Phase 1 | 6.7 (10.7) | 2.3 (4.9)
  Difference Post Phase 2 | -12 (10.5) | -5 (11.4)

2. Secondary Outcome: Change in Controlled Oral Word Association Test (COWA) Score
Description: This is a measure of attention, executive function, and word-retrieval. COWA scores range from 0 to infinity. Lower scores represent more language impairment.
Time Frame: Baseline, 1 week following each intervention period
Measure: Mean (Standard Deviation); unit: Number of Correct Items on COWA Test
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
Number of Correct Items on COWA Test
  Post Phase 1 | 6 (7.2) | 8 (11.3)
  Post Phase 2 | 3.7 (4.0) | 7.5 (10.6)

3. Secondary Outcome: Change in Quality of Sleep as Assessed by the Pittsburgh Sleep Quality Index (PSQI)
Description: Change in quality of sleep measured with The Pittsburgh Sleep Quality Index (PSQI). This has 7 items with each item scored from 0 to 3. Overall score ranges from 0 to 21 with higher scores representing poor sleep quality.
Time Frame: Baseline, 1 week following each intervention period and 8 weeks following both intervention periods
Measure: Mean (Standard Deviation); unit: Score on Pittsburgh Sleep Quality Index
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
Score on Pittsburgh Sleep Quality Index
  Difference Post Phase 1 | 0.67 (7.57) | 5.67 (5.51)
  Difference Post Phase 2 | -0.33 (2.89) | -3.33 (3.06)

4. Secondary Outcome: Change in Anxiety as Assessed by the State Trait Anxiety Inventory (STAI)
Description: Change in anxiety measured with State Trait Anxiety Inventory. This is a 40-item questionnaire scored on a 4 point likert scale (1-4). Overall score ranges from 40 to 160 with higher scores representing greater (worse) anxiety. STAI Part 1 Score range 20-80 and STAI Part 2 score range 20-80 with higher scores representing greater (worse) anxiety.
Time Frame: Baseline, 1 week following each intervention period and 8 weeks following both intervention periods
Population: Participants with data collected. One participant in each group was unable to complete this self-reported index due to the severity of their language deficits related to their aphasia prohibiting them from completing the questionnaire items.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 2 | 2
score on a scale
  Difference Post Phase 1, STAI Part 1 | 10 (9.9) | -4.5 (6.36)
  Difference Post Phase 2, STAI Part 1 | -7 (8.49) | 8.5 (2.12)
  Difference Post Phase 1, STAI Part 2 | -3.5 (0.71) | 1 (7.07)
  Difference Post Phase 2, STAI Part 2 | -0.5 (7.78) | 2 (2.83)

5. Secondary Outcome: Change in Sleep Medication Dosage
Description: Change in number of doses of sleep medication taken per week
Time Frame: Baseline, 1 week following each intervention period
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
mg
  Difference Post Phase 1 | 0 (0) | 0 (0)
  Difference Post Phase 2 | 0 (0) | 0 (0)

6. Secondary Outcome: Change in Sleep Medication Frequency
Description: Change in frequency of sleep medication taken per week.
Time Frame: Baseline, 1 week following each intervention period and 8 weeks following both intervention periods
Measure: Mean (Standard Deviation); unit: Number of Doses taken per week
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
Number of Doses taken per week
  Difference Post Phase 1 | 0 (0) | 0 (0)
  Difference Post Phase 2 | 0 (0) | 0 (0)

7. Secondary Outcome: Change in Absolute Power on EEG
Description: Measurement of brainwave activity (absolute power in microvolts) in each frequency band (alpha, beta, theta, delta, gamma) on Quantitative EEG (qEEG). The difference in average absolute power is combined to report all frequency bands.
Time Frame: Baseline, 1 week following each intervention period
Measure: Mean (Standard Deviation); unit: EEG Absolute Power (microvolts)
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
EEG Absolute Power (microvolts)
  Difference Post Phase 1 | 0.53 (0.66) | 0.42 (1.15)
  Difference Post Phase 2 | -0.49 (0.64) | 0.38 (0.34)

8. Secondary Outcome: Change in Peak Amplitude Frequency on EEG
Description: Measurement of brainwave activity (peak alpha amplitude frequency in hertz) on qEEG.
Time Frame: Baseline, 1 week following each intervention period
Measure: Mean (Standard Deviation); unit: Peak amplitude frequency (Hz)
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
Peak amplitude frequency (Hz)
  Difference Post Phase 1 | 0.29 (0.72) | 0.24 (0.11)
  Difference Post Phase 2 | 0.72 (0.71) | -0.04 (0.06)

9. Secondary Outcome: Change in EEG Absolute Power Z-scores
Description: Comparison of z-scores for absolute power pre- and post-interventions. A Z-score of 0 represents the population mean. A z-score of <-2 and >2 is clinically worse than values approximating the z score central value (0) the population mean.
Time Frame: Baseline, 1 week following each intervention period
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
z score
  Difference Post Phase 1 | 0.53 (0.29) | 0.23 (0.44)
  Difference Post Phase 2 | -0.41 (0.27) | 0.14 (0.05)

10. Secondary Outcome: Change in EEG Peak Amplitude Frequency Z-scores
Description: Comparison of z-scores for peak alpha amplitude frequency pre- and post-interventions. A z-score of <-2 and >2 is clinically worse than values approximating the z score central value (0) the population mean.
Time Frame: Baseline, 1 week following each intervention period
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
z score
  Difference Post Phase 1 | 0.34 (0.74) | 0.31 (0.14)
  Difference Post Phase 2 | 0.58 (0.7) | -0.07 (0.02)

11. Secondary Outcome: Change in EEG Coherence Z-scores
Description: Comparison of z-scores for coherence between EEG sites in each of the frequency bands (alpha, beta, theta, delta, gamma). A Z-score of 0 represents the population mean. A z-score of <-2 and >2 is clinically worse than values approximating the z score central value (0) the population mean. The difference in average z-score is combined to report coherence in all frequency bands.
Time Frame: Baseline, 1 week following each intervention period
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Active EEG Neurofeedback, Then Sham Neurofeedback | Sham Feedback, Then Active Neurofeedback
Number analyzed (Participants) | 3 | 3
z-score
  Difference Post Phase 1 | 0.13 (0.32) | -0.11 (0.31)
  Difference Post Phase 2 | -0.04 (1.02) | -0.09 (0.4)

ADVERSE EVENTS:
Time Frame: enrollment until end of follow up, approximately 5 weeks
Groups:
- Active EEG Neurofeedback: 15 sessions of active neurofeedback at a frequency of 3-5 sessions per week for a duration of 3-5 weeks .
Arm/Group | Active EEG Neurofeedback | Sham Feedback
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
This study was discontinued due to lack of funding before we could enroll our target number of participants and complete the study. Therefore, we couldn't complete the full analysis initially planned to determine the intervention's efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT04290988/Prot_SAP_000.pdf